CLINICAL TRIAL: NCT06865534
Title: Medical Students and Their Perception of Large Language Models (LLMs) in Gynecologic Oncology
Brief Title: Large Language Models to Aid Gynecological Oncology Treatment
Acronym: EASING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 25-29 ANZ; 25-29 ANZ (Other: Philipps University Marburg)
Record Dates: First submitted 2025-02-11; First posted 2025-03-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: large language models; clinical decision support; gynecological oncology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local language model first (Other): Group will be given access to local language model first after using ChatGPT
  Interventions: Other: Local language model
- Guideline pdf first (Other): Group will be given access to guideline pdf first after using ChatGPT
  Interventions: Other: Guideline pdf

INTERVENTIONS:
Other: Local language model — Group will be given access to local language model first after using ChatGPT and then will get access to pdf file
  Arms: Local language model first
Other: Guideline pdf — Group will be given access to pdf file after ChatGPT and then to a local language model
  Arms: Guideline pdf first

SUMMARY:
This trial aims to assess the impact of providing medical students with access to large language models, in comparison to treatment guideline pdfs, on treatment concordance with a conventional multidisciplinary tumor board

DETAILED DESCRIPTION:
Advanced artificial intelligence (AI) technologies, particularly large language models such as OpenAI's ChatGPT, hold significant potential for enhancing medical decision-making. While ChatGPT was not specifically designed for medical applications, it has shown utility in various healthcare scenarios, including answering patient inquiries, drafting medical documentation, and aiding clinical consultations. Despite these advancements, its role in supporting treatment decision-making-particularly in complex oncological cases-remains underexplored.

Treatment decision-making in gynecological oncology is a multifaceted process that integrates evidence-based guidelines, tumor biology, patient-specific factors, and clinical expertise. AI tools like ChatGPT could potentially assist in synthesizing relevant guideline-based recommendations, improving decision accuracy, and facilitating more efficient clinical workflows. However, ChatGPT is not specifically tailored for oncological treatment decisions and lacks comprehensive validation in this domain. Additionally, it may generate misinformation or plausible-sounding but inaccurate recommendations, which could impact clinical judgment. Therefore, understanding how medical professionals, including students and early-career physicians, interact with such AI tools is essential before broader integration into clinical practice. Locally deployable models, such as Llama, enable secure, on-premise usage while retrieval-augmented generation ensures guideline-compliant recommendations.

This study will investigate the impact of language models on treatment decision support for medical students managing gynecological oncology cases. This is a crossover study, where participants will be randomized into two groups. All participants begin with access to ChatGPT for two vignettes. They then proceed with two cases using either a locally deployed language model, followed by two cases relying on guideline PDFs, or vice versa.

Each participant will analyze clinical cases, propose treatment plans, and rate their confidence in their decisions and decision support system usability. This study aims to provide insights into the potential benefits and limitations of integrating AI tools like ChatGPT into oncological treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

- Medical students having started with clinical subjects

Exclusion Criteria:

- Not being a medical student

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment concordance with tumor board decisions | directly (within 10 minutes) after Intervention
  Participants in each group select treatment modalities for case vignettes

SECONDARY OUTCOMES:
Treatment confidence | directly (within 10 minutes) after Intervention
  For each case participants will be asked for their treatment confidence (VAS 0-10). The mean score will be compared between decision support groups.
Time spent for treatment decision | directly (within 10 minutes) after Intervention
  Time (in seconds) participants spend per case between the decision support groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Griewing, MD PhD, Principal Investigator — Philipps University Marburg
Locations (1):
- Institute for Digital Medicine, University Hospital of Giessen and Marburg, Philipps University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No